CLINICAL TRIAL: NCT02210507
Title: Beta-carotene Absorption and Bioconversion to Vitamin A in a Biofortified Cassava Gari Meal and a White Cassava Gari Meal With Added Red Palm Oil
Brief Title: Beta-carotene Absorption and Bioconversion to Vitamin A From Biofortified Cassava Gari
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: HarvestPlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FL93
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Vitamin A Deficiency
Keywords: vitamin A; retinol; carotenoids
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- White cassava gari (Experimental): A single meal containing 400 gm of garified non-biofortified (white) cassava with retinyl palmitate reference dose.
  Interventions: Other: White cassava gari
- White cassava gari + red palm oil (Experimental): A single meal containing 400 gm of garified non-biofortified (white) cassava with red palm oil.
  Interventions: Other: White cassava gari + red palm oil
- Biofortified cassava gari (Experimental): A single meal containing 400 gm of garified biofortified cassava.
  Interventions: Other: Biofortified cassava gari

INTERVENTIONS:
Other: Biofortified cassava gari — Cassava, bred to contain high amounts of vitamin A-forming carotenoids (primarily beta-carotene and its cis-derivatives).
  Arms: Biofortified cassava gari
Other: White cassava gari — Non-biofortified (white) cassava and a retinyl palmitate reference dose.
  Arms: White cassava gari
Other: White cassava gari + red palm oil — Non-biofortified (white) cassava gari containing red palm oil.
  Arms: White cassava gari + red palm oil

SUMMARY:
The goal of the research study is to determine the absorption, metabolism, and bioconversion of carotenoids such as beta-carotene to vitamin A from gari made with biofortified cassava compared to a mixture of red palm oil and gari made from typical white cassava.

DETAILED DESCRIPTION:
Vitamin A deficiency (VAD) is a major public health problem in most of the developing world, especially Southern Asia and Sub-Saharan Africa. The primary issue in vitamin A deficient populations is the low vitamin A content of the diet. Beta-carotene is the most abundant provitamin A carotenoid in nature and in human tissues. Increasing the concentrations of bioavailable vitamin A-forming carotenoids in staple foods by selective breeding is a good strategy for improving vitamin A status. Cassava, bred to contain high amounts of vitamin A-forming carotenoids is one such food, since it is a staple crop in Africa and parts of South America. A popular cassava product Africa is gari, which is fermented, dewatered, milled, and roasted so that it can be used for porridges and in baking. However, the effect of feeding biofortified gari meals on carotenoid and vitamin A concentrations in the body is not known. A common practice is to add red palm oil to typical white cassava gari. Red palm oil is a very rich source of alpha-carotene and beta-carotene, in highly bioavailable forms. Unfortunately, little is known of the bioconversion of red palm oil cassava mixture carotenoids to vitamin A.

The primary purpose of this study is to determine the effect of consuming gari that is made from biofortified cassava on carotenoid and vitamin A concentrations. The investigators will compare carotenoid and vitamin A concentrations in individuals fed biofortified gari to the same individuals fed gari made from ordinary cassava. The investigators hypothesis is that the biofortified gari will increase carotenoid and vitamin A concentrations in triacylglycerol-rich plasma (TRL). The secondary purpose of this study is to investigate the effect of a meal of high carotenoid red palm oil added to typical white gari on carotenoids and vitamin A. Adding red palm oil to white gari should be an effective method for increasing carotenoids and vitamin A status in the gari meal, and thus humans. The investigators will match the amount of retinol equivalents in the biofortified cassava gari and red palm oil-containing white cassava gari. This will let us compare their effectiveness at increasing carotenoid and vitamin A concentrations in the TRL plasma fraction after consumption. This will allow us to compare their bioavailability and bioconversion efficiencies.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-pregnant, non-lactating
* premenopausal women
* non-smoking
* body mass index between 18 and 35
* total cholesterol concentrations between 90 and 225 mg/dL
* blood pressure under 140/90 mm Hg

Exclusion Criteria:

* anemia, Hemoglobin less than 11.5 g/dL
* medications such as gemfibrozil, niacin, lovastatin, simvastatin, ezetimibe)
* medications that affect retinoid or carotenoid metabolism (Accutane)
* medications that impair fat absorption (Xenical, orlistat)
* dietary supplements containing vitamin A

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in vitamin A in triacylglycerol-rich lipoprotein (TRL) fraction of plasma | 2, 3.5, 5, 7.25, and 9.5 hours after a meal
  Vitamin A is measured by standard methods involving ultracentrifugation (to concentrate the TRL fraction) followed by reversed-phase high pressure liquid chromatography (HPLC) using electrochemical detection.

SECONDARY OUTCOMES:
Change in carotenoids in triacylglycerol-rich lipoprotein (TRL) fraction of plasma | 2, 3.5, 5, 7.25, and 9.5 hours after a meal
  Carotenoids will be measured by standard methods involving ultracentrifugation (to concentrate the TRL fraction) followed by reversed-phase HPLC using electrochemical detection.

CONTACTS AND LOCATIONS:
Overall Officials: Betty J Burri, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- See also: USDA, ARS, WHNRC — http://www.ars.usda.gov/Main/docs.htm?docid=11240